CLINICAL TRIAL: NCT04753216
Title: A Phase II Trial of Irinotecan Liposome and Bevacizumab in Women With Platinum Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Irinotecan Liposome and Bevacizumab for the Treatment of Platinum Resistant, Recurrent, or Refractory Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ipsen (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniela Matei, Daniela Matei, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 20G02; STU00213582 (CTRP (Clinical Trial Reporting Program)); NU 20G02 (Other: Northwestern University); P30CA060553 (NIH); NCI-2021-00765 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Refractory Fallopian Tube Carcinoma; Refractory Ovarian Carcinoma; Refractory Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (bevacizumab, irinotecan sucrosofate) (Experimental): Patients receive bevacizumab IV and irinotecan sucrosofate IV over 90 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Irinotecan Sucrosofate

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Drug: Irinotecan Sucrosofate — Given IV
  Other Names: Irinotecan Liposome; MM-398; nal-IRI; Nanoliposomal Irinotecan; Nanoparticle Liposome Formulation of Irinotecan; Onivyde; PEP02

SUMMARY:
This phase II trial investigates the effect of irinotecan liposome and bevacizumab in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that shows less response to platinum therapy (platinum resistant), has come back (recurrent), or does not respond to treatment (refractory). Irinotecan liposome may help block the formation of growths that may become cancer. Bevacizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving irinotecan liposome and bevacizumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the antineoplastic efficacy of irinotecan sucrosofate (irinotecan liposome) in combination with bevacizumab in women with recurrent, platinum resistant ovarian cancer, as measured by the objective response rate (ORR).

SECONDARY EFFICACY OBJECTIVES:

I. To determine the overall best response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in women with recurrent, platinum resistant ovarian cancer who have received treatment with irinotecan liposome in combination with bevacizumab.

II. To determine the clinical benefit rate (CBR) for irinotecan liposome in combination with bevacizumab in women with recurrent, platinum resistant ovarian cancer.

III. To calculate the duration of response (DOR) for irinotecan liposome in combination with bevacizumab in women with recurrent, platinum resistant ovarian cancer.

IV. To calculate the duration of stable disease (duration of SD) for irinotecan liposome in combination with bevacizumab in women with recurrent, platinum resistant ovarian cancer.

V. To calculate the time to response (TTR) for irinotecan liposome in combination with bevacizumab in women with recurrent, platinum resistant ovarian cancer.

VI. To measure median progression-free survival (PFS) in women with recurrent, platinum resistant ovarian cancer who have received treatment with irinotecan liposome in combination with bevacizumab.

VII. To measure 16 week progression-free survival (PFS-16) in women with recurrent, platinum resistant ovarian cancer who have received treatment with irinotecan liposome in combination with bevacizumab.

SECONDARY SAFETY OBJECTIVE:

I. To assess the toxicity profile of irinotecan liposome in combination with bevacizumab in women with recurrent, platinum resistant ovarian cancer according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

OUTLINE:

Patients receive bevacizumab intravenously (IV) and irinotecan sucrosofate IV over 90 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.

  * NOTE: Subjects with carcinosarcoma histology and/or mixed epithelial histology are not eligible.
* Subjects must have recurrent, platinum resistant or refractory disease, defined as progression < 6 months after completion of a platinum-based chemotherapy regimen or as persistent disease that remains after completion of a platinum-based therapy
* Subjects must have measurable disease as assessed by RECIST 1.1
* Subjects must have received at least 1 but no more than 3 prior platinum-based chemotherapy regimens
* Subjects must have adequately recovered (in the opinion of the treating investigator) from adverse events due to prior anti-cancer therapy, with the exceptions of any grade alopecia and =< grade 2 peripheral neuropathy per NCI-CTCAE version 5.0
* Subjects must be age >= 18 years
* Subjects must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Hemoglobin >= 9.0 g/dL (within =< 28 days prior to registration)
* White blood cell (WBC) count >= 3.0 x 10^9/L (within =< 28 days prior to registration)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within =< 28 days prior to registration)
* Platelet count >= 75 x 10^9/L (within =< 28 days prior to registration)
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SPGT]) =< 2.5 x ULN or =< 5.0 x ULN for subjects with liver metastases
* Serum albumin >= 3.0 g/dL
* Serum creatinine =< 1.5 x ULN
* Urine protein < 2+ (urine dipstick) or < 100 mg/dL (random protein urinalysis) or < 1 g/24h (24 hour urine collection)
* International normalized ratio (INR) =< 1.5 x ULN or for subjects receiving anticoagulant therapy, INR must be within the therapeutic range of intended use of anticoagulants, as determined by the treating investigator
* Activated partial thromboplastin Time (aPTT) =< 1.5 x ULN or for subjects receiving anticoagulant therapy, aPTT must be within the therapeutic range of intended use of anticoagulants, as determined by the treating investigator
* For subjects with a known history of human immunodeficiency virus (HIV), the HIV viral load must be undetectable for >= 6 months prior to registration, and subjects must be receiving effective anti-retroviral HIV therapy, if indicated

  * NOTE: HIV testing is not required for subjects without a known history of HIV, unless mandated by a local health authority
* For subjects with a known history of hepatitis B virus (HBV) infection or hepatitis C virus (HCV) infection, the HBV/HCV viral load must be undetectable, and subjects must be receiving effective suppressive HBV/HCV therapy, if indicated.

  * NOTE: HBV and HCV testing is not required for subjects without a known history of HBV or HCV, unless mandated by a local health authority
* Subjects with previously treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for >= 28 days prior to registration, and any neurologic symptoms have returned to baseline
* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen for this trial are eligible
* Subjects with a known history severe cardiac disease, current symptoms of cardiac disease (e.g., unstable angina pectoris or cardiac arrhythmia), or a history of treatment with cardiotoxic agents should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, these subjects must be class 2B or better
* For subjects with hypertension, hypertension must be well controlled on medication.

  * NOTE: Uncontrolled hypertension is defined as a consistent blood pressure (bp) of >= 160 mmHg systolic or >= 100 mmHg diastolic, on initial and repeat checks
* Females of reproductive potential must agree to undergo a urine or serum pregnancy test, and the results must be negative in order to initiate treatment.

  * NOTE: A female of reproductive potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Females of reproductive potential must agree to use adequate contraception (abstinence or two methods of birth control, such as a barrier method in combination with hormonal contraception) while receiving trial therapy and for 6 months following completion of trial therapy. Should a woman become pregnant or suspect she is pregnant while is participating in this study, she should inform her treating physician immediately.

  * NOTE: A female of reproductive potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Subjects must agree to not nurse/breastfeed while receiving trial therapy and for 6 months after the last dose of trial therapy.

  * Note: These subjects are excluded because there is an unknown but potential risk for adverse events to the nursing infant
* Surgical wounds (including wounds from tooth extractions and jaw-invasive dental procedures) must be fully healed and subjects must have adequately recovered (in the opinion of the treating investigator) from adverse events due to prior surgical procedures
* Subjects (or their legally authorized representative if subject has impaired decision-making capacity) must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Exclusions for receipt of prior systemic anti-cancer therapy:

  * Subjects must not have received any prior irinotecan-based therapies.
  * Subjects must not have received more than 3 prior platinum-based chemotherapy regimens.
  * Subjects must not have received more than 2 prior non-platinum, cytotoxic chemotherapy regimens.
  * Note: Prior receipt of non-VEGF-targeting biological therapies is permitted. These may include but are not limited to hormonal therapies, immunotherapies, monoclonal antibodies (mAbs), tyrosine kinase inhibitors (TKIs), poly (ADP-ribose) polymerase (PARP) inhibitors, or other targeted agents. Refer to the below exclusion criterion for washout rules
* Exclusions for washout from prior systemic anti-cancer therapy:

  * Subjects must not have received chemotherapy, immunotherapy, monoclonal antibody (mAb) therapy, hormonal therapy, or other targeted therapy within =< 14 days prior to registration.
  * Subjects must not have received investigational agents or investigational devices within =< 14 days prior to registration.
  * Subjects must not have received VEGF-targeting agents, including bevacizumab, within =< 6 months prior to registration
* Subjects must not have received prior radiotherapy to the pelvis or abdomen within =< 3 months prior to registration. Subjects must not have received prior radiotherapy to other areas within =< 14 days prior to registration
* Subjects must not have undergone a surgical procedure or jaw-invasive dental procedure (including tooth extraction) within =< 28 days prior to registration
* Subjects must not have a known history of hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, irinotecan liposome, or any of their excipients
* Subjects must not have received hematologic growth factors and/or blood products (transfusions) within =< 28 days prior to registration
* Subjects must not be taking any of the medications listed as prohibited medications and therapies. Subjects receiving any medications or substances that are known strong CYP3A4 inducers, known strong CYP3A4 inhibitors, and/or known strong UGT1A1 inhibitors are ineligible.

  * Known strong CYP3A4 inducers must be discontinued at least 2 weeks prior to initiation of irinotecan liposome to be eligible.

    * Strong CYP3A4 inducers include, but are not limited to, the following: phenytoin, phenobarbital, primidone, carbamazepine, rifampin, rifabutin and rifapentine.
  * Known strong CYP3A4 and UGT1A1 inhibitors must be discontinued at least 1 week prior to initiation of irinotecan liposome to be eligible.

    * Strong CYP3A4 inhibitors include, but are not limited to, the following: ketoconazole, clarithromycin, indinavir, itraconazole, lopinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telaprevir, voriconazole. (Note: fosaprepitant is permitted).
    * Strong UGT1A1 inhibitors include, but are not limited to, the following: atazanavir, gemfibrozil, indinavir and ketoconazole
  * NOTE: Sites should refer to a current pharmacy reference manual for a full list of strong CYP3A4 inducers/inhibitors and strong UGTA1 inhibitors
* Subjects must not have active peptic ulcer disease, active inflammatory bowel disease, active ulcerative colitis, or other active gastrointestinal condition with increased risk of perforation. Subjects must not have a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within =< 6 months prior to registration
* Subjects must not have a history of bowel obstruction within =< 6 months prior to registration. Subjects also must not have:

  * Current evidence of tumor recto-sigmoid involvement by pelvic examination
  * Current tumor bowel involvement on computed tomography (CT) scan
  * Current clinical symptoms of bowel obstruction
* Subjects must not have a history of a significant thromboembolic or vascular disorders within =< 3 months prior to registration, including but not limited to:

  * Pulmonary embolism
  * Deep vein thrombosis
  * Other arterial or venous thromboembolic events
  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Peripheral arterial ischemia >= grade 3 (per NCI-CTCAE v5.0)
* Subjects must not have a history of a significant bleeding disorder within =< 6 months prior to registration, including but not limited to:

  * Hematemesis, hematochezia, melena or other gastrointestinal bleeding >= grade 2 (per NCI-CTCAE v5.0)
  * Hemoptysis of 1/2 teaspoon (2.5 mL) or more of red blood, or other pulmonary bleeding >= grade 2 (per NCI-CTCAE v5.0)
  * Hematuria or other genitourinary bleeding >= grade 2 (per NCI-CTCAE v5.0)
* Subjects must not have a current non-healing wound, bone fracture, skin ulcer, or osteonecrosis of the jaw
* Subjects must not be pregnant or expecting to conceive from the time of informed consent through 6 months after the last dose of trial treatment.

  * NOTE: These subjects are excluded because there is an unknown but potential risk for adverse events to the developing fetus
* Subjects must not have a known UGT1A1* variant or Gilbert's syndrome
* Subjects must not have received a live vaccine within =< 30 days prior to registration.

  * NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines and are not allowed
* Subjects must not have a condition or an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Ongoing or active infection requiring systemic treatment, except uncomplicated urinary tract infection (UTI) or uncomplicated upper respiratory tract infection (URI);
  * Psychiatric illness/social situation that would limit compliance with study requirements;
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the subject's safety or study endpoints

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela E Matei, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Screening - 1st Response Assessment
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Started | 3
Cycle 1 | 3
Cycle 2 | 3
1st Response Assessment | 2
Completed | 2
Not Completed | 1
Not completed — Adverse Event | 1
Period: Cycle 3 - 2nd Response Assessment
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Started | 2
Cycle 3 | 2
Cycle 4 | 2
2nd Response Assessment | 2
Completed | 1
Not Completed | 1
Not completed — Disease Progression | 1
Period: Cycle 5 - 3rd Response Assessment
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Started | 1
Cycle 5 | 1
Cycle 6 | 1
3rd Response Assessment | 0
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Survival Follow-Up
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  40-49 | 1
  60-69 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Defined as the proportion of treated subjects who experience an objective response, confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
  Complete Response (CR) = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR) = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD) = Neither sufficient shrinkage to qualify
Time Frame: Up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 2
Participants
  Partial Response | 2
  Complete Response | 0

2. Secondary Outcome: Overall Best Response
Description: Will tabulate the proportion of subjects who experience each the following as their best response to trial therapy: CR, PR, stable disease (SD), progressive disease (PD) or not evaluable (NE) per RECIST 1.1.
  Complete Response (CR) = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR) = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD) = Neither sufficient shrinkage to qualify
Time Frame: Approximately 29 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 2
Participants
  Stable Disease | 0
  Progressive Disease | 0
  Partial Response | 2
  Complete Response | 0

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: To determine the CBR, this endpoint will calculate the proportion of treated, evaluable subjects who experience clinical benefit from trial therapy. Clinical benefit is defined as confirmed complete response (CR); confirmed partial response (PR); or stable disease (SD) for ≥ 4 months (calculated from the initiation of trial therapy on C1D1) per RECIST 1.1.16. Will tabulate the proportion of subjects who experience each of the following as their best response to trial therapy: CR, PR, stable disease (SD), progressive disease (PD) or not evaluable (NE) per RECIST 1.1. CBR data will be collected from baseline until the subject experiences disease progression initiates subsequent anti-cancer therapy, or completes study participation (whichever occurs first).
Time Frame: Approximately 29 Weeks
Measure: Number; unit: Participants
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 2
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: To calculate the DOR for the combination of irinotecan liposome and bevacizumab, this endpoint will be calculated as the time that elapsed between the day of first documented response to trial therapy (CR or PR, whichever is first recorded) and subsequent disease progression (taking as reference for progressive disease the smallest tumor measurements recorded on study). For DOR analysis, response is defined as complete response (CR) or partial response (PR) per RECIST 1.1; and disease progression is defined as progressive disease (PD) per RECIST 1.1.16 DOR data will be collected from the time of first response to trial therapy until the subject experiences disease progression, initiates subsequent anti-cancer therapy, or completes study participation (whichever occurs first). If disease progression is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the DOR will be censored as the last available disease assessment.
Time Frame: Approximately 29 Weeks
Population: 1 patient had PR and then progressed without a subsequent scan and is not included in number of evaluable patients
Measure: Number; unit: Weeks
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 1
Weeks | 9.5

5. Secondary Outcome: Duration of Stable Disease
Description: To calculate the Duration of SD (CR, PR, and SD) for the combination of irinotecan liposome and bevacizumab, this endpoint will be calculated as the time that elapsed between the day of initiation of trial therapy and subsequent disease progression (taking as reference for progressive disease the smallest measurements recorded on study). Duration of SD analysis will capture subjects who achieve a best response of CR, PR, or SD, as defined per RECIST 1.1. For Duration of SD analysis, disease progression is defined as progressive disease (PD) per RECIST 1.1. Duration of SD data will be collected from baseline until the subject experiences disease progression, initiates subsequent anti-cancer therapy, or completes study participation. If disease progression is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the Duration of SD will be censored as the last available disease assessment.
Time Frame: Approximately 29 Weeks
Measure: Number; unit: weeks
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 1
weeks | 14

6. Secondary Outcome: Time to Response (TTR)
Description: For TTR analysis, a response to therapy is defined as a confirmed complete response (CR) or confirmed partial response (PR) per RECIST 1.1.
Time Frame: Approximately 29 Weeks
Measure: Number; unit: days
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 2
days
  Pt 01-01-101 | 137
  Pt 01-01-102 | 80

7. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: This endpoint will calculate the progression-free survival time as the time that elapsed between the initiation of trial therapy (C1D1) and the day of first documented disease progression or death from any cause for all evaluable subjects. Per RECIST 1.1, Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Approximately 29 Weeks
Measure: Number; unit: Days
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 1
Days | 117

8. Secondary Outcome: Progression Free Survival
Description: This endpoint will be calculated based on the proportion of subjects who are alive and progression-free at 16 weeks after initiating trial therapy.
  Per RECIST 1.1, Progressive Disease (PD) = At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: At 16 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 2
participants | 1

9. Secondary Outcome: Number of Observed Serious and Other (Not Including Serious) Adverse Events
Description: Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events 5.0 (NCI-CTCAE v5.0).
Time Frame: Approximately 29 Weeks
Measure: Number; unit: Adverse Events
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
Number analyzed (Participants) | 3
Adverse Events | 107

ADVERSE EVENTS:
Time Frame: All routine AEs, regardless of attribution or clinical significance, occurring from the time of subject registration, through 30 days after the last administration of trial therapy, must be recorded. Any event that occurs more than 30 days after the last dose of trial therapy and is attributed (possibly, probably, or definitely) to the agent(s) must also be reported as an adverse event or expedited adverse event, as applicable. This took place over a 29 week period.
Description: An adverse event is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product or undergoing an experimental intervention, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product or experimental intervention.
Arm/Group | Treatment (Bevacizumab, Irinotecan Sucrosofate)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab, Irinotecan Sucrosofate) (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab, Irinotecan Sucrosofate) (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 1 (10)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (7)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (8)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (7)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (6)
Nausea (Gastrointestinal disorders) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (7)
Platelet count decreased (Investigations) | 1 (6)
Proteinuria (Renal and urinary disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT04753216/Prot_SAP_001.pdf